CLINICAL TRIAL: NCT06491628
Title: Liver Function Abnormalities in Patients With Acute Heart Failure in Sohag University Hospitals
Brief Title: Liver Function Abnormalities in Patients With Acute Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Saber, Liver function abnormalities in patients with acute heart failure in Sohag University Hospitals, Sohag University
Other Study IDs: LFTs abnormalities in AHF
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Acute Heart Failure
Keywords: LFTs, AHF
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Acute decompensated heart failure (de novo or as decompensation of chronic heart failure): This umbrella term includes patients presenting forthe first time with typical symptoms and signs of heart failure(de novo AHF) and also those with worsening of their pre-existing cardiomyopathy (acute decompensated heart failure).
  Interventions: Behavioral: Avoiding the risk factors
- Pulmonary edema: It's the real clinical presentation of AHF, typically, signs and symptoms develope rapidly and patients demonstrate severe respiratory distress with tachypnea, orthopnea and pulmonary congestion
  Interventions: Behavioral: Avoiding the risk factors
- Hypertensive acute heart failure: the condition is associated with elevated blood pressure with accompanying dyspnea. orthopnea and pulmonary congestion, often in patients with relatively preserved left ventricle ejection fraction
  Interventions: Behavioral: Avoiding the risk factors
- cardiogenic shock: severe peripheral hypoperfusion wih subsequent end organs damage,typically it's associated with low blood pressure and low urine output
  Interventions: Behavioral: Avoiding the risk factors
- Acute coronary syndrome complicated by heart failure: characterized by complex structural, hemodynamic and neurohormonal interaction need urgent referral for coronary intervention poor outcome
  Interventions: Behavioral: Avoiding the risk factors

INTERVENTIONS:
Behavioral: Avoiding the risk factors — Exercise, Salt and lipid reduction in diet, smoking cessation

SUMMARY:
The aim of this study is to evaluate liver function test abnormalities and to identify associated cardiac and non cardiac factors mediating hepatic impairment in acute heart failure patients

DETAILED DESCRIPTION:
Cardiac failure has a negative impact on the function of all parenchymatous organs, based both on the low organ perfusion in the left-sided failure and on the venous congestion in the right-sided failure.

The pathophysiology of acute heart failure (AHF) is complex and not fully understood. It has been hypothesized that an episode of acute decompensation affects not only the cardiovascular system itself, but may also deteriorate the function of other organs, c ausing serious clinical consequences. Liver involvement has been mostly described and investigated in patients with chronic HF.

Liver enzyme alterations are usually classified as relating predominantly to liver cell necrosis (signified by transaminase elevations) or predominantly to cholestasis (signified by elevated alkaline phosphatase (AP) level).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 yrs or older presenting with AHF

Exclusion Criteria:

* Congenital heart disease
* acute and chronic liver diseases

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged 18 yrs or older presenting with AHF
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Liver function abnormalities in patients with acute heart failure in Sohag University Hospitals | baseline
  assessment the LFTs abnormalities and factors mediating hepatic impairment in patients with AHF

SECONDARY OUTCOMES:
Liver function abnormalities in patients with acute heart failure in Sohag University Hospitals | 1 year
  assessment the LFTs abnormalities and factors mediating hepatic impairment in patients with AHF

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Saad, Study Chair — Sohag University; Haitham Mohammad, Study Chair — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt